CLINICAL TRIAL: NCT00974909
Title: Percutaneous Tibial Nerve Stimulation in the Treatment of Fecal Incontinence: a Multi-center, Randomized, Placebo Controlled Study
Brief Title: Percutaneous Tibial Nerve Stimulation in the Treatment of Fecal Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-2-079; NL 28955.068.09; MEC 09-2-079
Record Dates: First submitted 2009-09-08; First posted 2009-09-11 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2010-09

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Active Comparator): Treatment group
  Interventions: Device: Urgent PC neuromodulation system
- sham group (Sham Comparator): Sham group
  Interventions: Device: Urgent PC neuromodulation system

INTERVENTIONS:
Device: Urgent PC neuromodulation system — Urgent PC neuromodulation system
  Arms: Treatment group
Device: Urgent PC neuromodulation system — Urgent PC neuromodulation system (sham)
  Arms: sham group

SUMMARY:
Background of the study:

Fecal incontinence is a complex problem. The social consequences of this problem result in a lower quality of life. The exact prevalence of FI is unknown, literature reports vary from 13-19%. There are variable treatment options depending on the patient and the etiology of the FI. Dietary manipulation, pharmacological intervention, pelvic floor physiotherapy, as well as surgical interventions are currently used to treat FI.

A promising current treatment is Percutaneous Tibial Nerve Stimulation (PTNS). The nerves in the spine that control bowel function also have branches which go to the ankle. Stimulating these nerves in the ankle has shown to be an effective treatment for FI in the short-term. The treatment has been shown to be safe and well tolerated by subjects with almost no morbidity in prior urology trials.

Objective of the study:

The objective of this study is to show that the results of PTNS are based on the treatment of electrical stimulation and not on a placebo effect with a sham treatment.

Study design:

This study is a multicenter, single-blinded, randomized, placebo-controlled trial.

Primary study parameters/outcome of the study:

The percentage of patients experiencing a ≥ 50% decrease in incontinence episodes from baseline after 9 weeks of treatment.

Secondary study parameters/outcome of the study (if applicable):

Mean change in the Cleveland Clinic Florida Fecal Incontinence Score (CCF-FI Score)

Mean change in Quality of Life scores in validated QoL questionnaires (SF-36, Digestive Health Status Instrument (DHSI), and Fecal Incontinence Quality of life)

Subject's and Physician's Global Impression

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Must be at least 18 years of age
* Fecal incontinence with solid or liquid stool causing disruption of the subject's lifestyle
* Psychological stability as determined by treating physician
* Willingness to commit to a rigid follow-up schedule and comply with the investigational plan
* Failed conservative therapy (i.e. dietary and behavioural modification, biofeedback techniques and exercises for pelvic floor muscle retraining)
* During treatment the patient exhibits an adequate motor and/or sensory response (flexion of toe and/or twinkling sensation)
* Is able to read and write

Exclusion Criteria:

* Major internal and/or external sphincter defect (defined as >33% of the anal circumference)
* Fecal impaction
* Pacemaker, implanted defibrillator
* Pregnancy or intention to become pregnant
* Neurogenic or congenital disorders resulting in FI
* Inability to travel to the clinic twice a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The percentage of patients experiencing a ≥ 50% decrease in incontinence episodes from baseline after 9 weeks of treatment and at six and twelve months follow-up. | 9 weeks

SECONDARY OUTCOMES:
Mean change in the Cleveland Clinic Florida Fecal Incontinence Score (CCF-FI Score) at 6 weeks and 9 weeks of treatment and at six and twelve months follow-up. | one year
Mean change in Quality of Life scores in validated QoL questionnaires (SF-36, Digestive Health Status Instrument (DHSI), and Fecal Incontinence Quality of life) at 6 weeks and 9 weeks of treatment and at six and twelve months follow-up. | one year
Subject's and Physician's Global Impression at 6 weeks and 9 weeks of treatment and at six and twelve months follow-up. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Baeten, prof phd md, Principal Investigator — Maastricht University Medical Center
Locations (3):
- CCDE - IMAD - Hôtel-Dieu, Nantes, France
- Università degli Studi di Roma "La Sapienza", Roma, Italy
- Maastricht university medical center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van der Wilt AA, Giuliani G, Kubis C, van Wunnik BPW, Ferreira I, Breukink SO, Lehur PA, La Torre F, Baeten CGMI. Randomized clinical trial of percutaneous tibial nerve stimulation versus sham electrical stimulation in patients with faecal incontinence. Br J Surg. 2017 Aug;104(9):1167-1176. doi: 10.1002/bjs.10590. PMID 28703936